CLINICAL TRIAL: NCT03777670
Title: Detecting Neonatal Sepsis by Immune-Metabolic Network Analysis
Brief Title: nSeP: Detecting Neonatal Sepsis by Immune-Metabolic Network Analysis
Acronym: nSeP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: Cardiff University (Other)
Responsible Party: Principal Investigator, Mallinath Chakraborty, Consultant in Neonatal Medicine, Cardiff and Vale University Health Board
Other Study IDs: 248404
Record Dates: First submitted 2018-12-13; First posted 2018-12-17 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Sepsis
Keywords: Newborn
MeSH Terms: conditions — Sepsis | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — RNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Infants with suspected sepsis
  Interventions: Diagnostic Test: Blood test
- Controls: Infants with no suspicion of sepsis
  Interventions: Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Blood test — Drop of blood for RNA and metabolic analysis

SUMMARY:
Diagnosis of neonatal sepsis remains a challenge due to non-specific signs and diagnostic inaccuracies. Studies have shown that this could lead to overdiagnosis and overuse of antibiotic treatment, with potential long-term adverse effects.

A systems approach towards diagnosing neonatal sepsis has been shown to have high accuracy in initial studies. This study aims to recruit a large validation cohort to confirm findings.

DETAILED DESCRIPTION:
Several studies have shown that changes in host gene expression may occur pre- symptomatically in response to infection in any part of the body, with the continuous interaction between blood and tissue allowing blood cells to act as biosensors for the changes (Manger and Relman, 2000, Liew et al., 2006). Genome wide analysis reveals coordinate expression that develop networks causally linked through pathways.

Earlier studies from our group investigating optimal methods for the sampling and extraction of neonatal whole transcription products (RNA) demonstrated the first feasibility studies for using genome wide RNA analysis as a methodological approach for identifying host biomarkers of infection and vaccination in early life (Smith et al., 2007, Flanagan et al., 2013). The sampling methods were further refined in 2015 with the development of a single drop methodology that has been extensively tested in a wide range of settings including the collection of neonatal samples in the home, at the point of Guthrie testing by mid-wives. Details of these methods have been recently submitted to the Nature Protocols journal. Further, we conducted early on virtual clinical trials using a super computing framework that simulated several 100,000 neonatal whole blood samples for predicting infection (Khondoker et al., 2010). Those investigations showed the requirement for multiple markers and ideally in discrete biological pathways underpinning causality (Khondoker et al., 2010, Watterson and Ghazal, 2010). Those investigations provided a strong foundation for initiating a case-control of neonatal sepsis (Dickinson et al., 2015). Accordingly, we were the first group to publish studies investigating the systemic immune response in neonates to sepsis by measuring the activity of all known human genes (Smith et al Nature comm. 2014). These computationally intensive investigations led to uncovering, for the first time, the pathway biology underlying neonatal sepsis with blood samples taken at the first clinical signs of suspecting an infection. A combination of machine learning, statistical and deep pathway biology analyses led to the identification of a 52-gene panel of biologically connected network modules. The modules comprise three central pathways, innate-immune or inflammatory, adaptive-immune and unexpectedly metabolic. The expression levels of particular combinations of biomarkers, and specifically those of a pathway previously unconnected to immune responses, gives an unusually high diagnostic quality. Despite patient heterogeneity, the 52-node dual biomarker network had greater than 99% accuracy for detecting bacterial infection with 100% sensitivity showing superior performance to previously characterised markers. Furthermore, these specific combinations of biomarkers allowed the detection of neonatal sepsis in samples which had displayed blood-culture negative results, illustrating the specific diagnostic benefits of the particular combinations of biomarkers. The unexpectedly high accuracy and sensitivity values could not have resulted from the investigation of any of the individual biomarkers alone, nor could they have been predicted. A critical part of these findings is the requirement of metabolic pathways for increasing both sensitivity and specificity. A subset of the metabolic markers encompass ligands (specifically small and medium chain fatty acids) that are derived from microbial metabolism, in particular from commensals and which are reflected in the faecal microbiome. To date these studies provide a proof of concept but need independent confirmatory studies as well as investigating specificity against non-bacterial (viral and fungal) infections and sterile inflammation. The urgent unmet medical question is whether predictive host pathways of infection can be used to first identify whether a patient is infected at or before clinical presentation and, to further discriminate between the type of infection (in particular bacterial or viral) and predictability of sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Screened with traditional tests (full-blood count [FBC], inflammatory markers like C-reactive protein [CRP], and blood-culture) for suspected sepsis (including non-infective inflammatory conditions) and started on antibiotics - potential cases.
* Being sampled for non-septic conditions (bloods sampling for routine monitoring, jaundice, hypoglycaemia, etc.) - controls.
* Informed consent from parents to use blood and stool samples (initial sample and 24-hour sample) and clinical data for study.

Exclusion Criteria:

* Language and communication issues, which will make it difficult to explain study and request informed consent.
* When an infant has a high chance of mortality in the next 24-hours.

Max Age: 4 Months | Sex: All
Age Groups: Child
Study Population: Newborn infants in the neonatal unit with a suspicion of sepsis
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Sepsis | 5-years
  Immune signature of sepsis

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Wales, Cardiff, South Glamorgan, United Kingdom

REFERENCES:
- [Derived] Chakraborty M, Rodrigues PRS, Watkins WJ, Hayward A, Sharma A, Hayward R, Smit E, Jones R, Goel N, Asokkumar A, Calvert J, Odd D, Morris I, Doherty C, Elliott S, Strang A, Andrews R, Zaher S, Sharma S, Bell S, Oruganti S, Smith C, Orme J, Edkins S, Craigon M, White D, Dantoft W, Davies LC, Moet L, McLaren JE, Clarkstone S, Watson GL, Hood K, Kotecha S, Morgan BP, O'Donnell VB, Ghazal P. nSeP: immune and metabolic biomarkers for early detection of neonatal sepsis-protocol for a prospective multicohort study. BMJ Open. 2021 Dec 30;11(12):e050100. doi: 10.1136/bmjopen-2021-050100. PMID 37010923